CLINICAL TRIAL: NCT02464709
Title: Daylight Mediated Photodynamic Therapy for Actinic Keratoses: a Multicentre Study Comparing Two Photosensitizers (BF-200 ALA Versus MAL)
Brief Title: Daylight PDT for Actinic Keratoses: a Multicentre Study Comparing Two Photosensitizers (BF-200 ALA Versus MAL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Päijänne Tavastia Central Hospital (Other); Tampere University Hospital (Other); Vaasa Central Hospital, Vaasa, Finland (Other); Tampere University (Other); STUK - Radiation and Nuclear Safety Authority: Finland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Q282dnro3/2015
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Actinic Keratosis; Natural Daylight Photodynamic Therapy
Keywords: Actinic Keratosis; Photodynamic Therapy; Natural Daylight
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; BF-200 ALA; methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Actinic keratosis patients (Experimental): Participant's AKs in facial skin or scalp are first clinically graded and demarcated in two symmetric treatment areas on different sides of face. The areas will be curettaged thinly and next a SPF20 sun protection cream is applied on all sun-exposed areas of the skin. Then a 0,25mm-thick layer of BF-200 ALA (aminolevulinic acid) gel is applied on one treatment side and MAL (methyl 5-aminolevulinate) cream on the other side. The sides will be randomized and the participant doesn't know which side is treated with which light sensitizer. After appropriate absorption time of 30 minutes the patients will be taken to the hospital balcony or yard for 2 hour illumination with natural daylight to accomplish the phototoxic reaction. Maximum dosage of light sensitizer will be 2 grams.
  Interventions: Drug: Aminolevulinic Acid; Drug: Methyl 5-aminolevulinate

INTERVENTIONS:
Drug: Aminolevulinic Acid — A 0,25mm-thick layer of BF-200 ALA (aminolevulinic acid, Ameluz®) light sensitizer gel is applied on one randomized treatment side of face.
  Other Names: BF-200 ALA; Ameluz®
Drug: Methyl 5-aminolevulinate — A 0,25mm-thick layer of MAL (methyl 5-aminolevulinate, Metvix®) light sensitizer cream is applied on one randomized treatment side of face.
  Other Names: MAL; Metvix®

SUMMARY:
This study compares two photosensitizing creams' BF-200 ALA's (aminolevulinic acid, Ameluz®) and MAL's (methyl 5-aminolevulinate, Metvix®) efficacy on actinic keratoses in natural daylight photodynamic therapy (NDL-PDT). The participants' facial skin or scalp will be randomized in two sides and one side is treated with BF-200 ALA and the other side with MAL. Result of the treatment is assessed with clinical examination 12 months after treatment. The investigators will also compare delayed skin reactions after treatment and cost-effectiveness of both photosensitizer creams.

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) is a widely used method in dermatology clinics for treatment of superficial skin cancers and premalignant lesions. Actinic keratoses (AKs) are premalignant skin lesions which develop due to long-lasting sun exposure and in time can progress into squamocellular skin cancer if left untreated. The incidence of AKs and skin cancers is rapidly booming as the elderly population increases in western countries. It is crucial to treat AKs early and effectively considering their tendency to progress into malign cancer. The current general consensus for treating AKs is to treat large sun-damaged skin areas simultaneously instead of separate AK lesions. Term "skin field cancerization" refers to presence of different degrees of visible and invisible dysplastic changes in widely sun-damaged skin. Natural daylight mediated photodynamic therapy (NDL-PDT) is a well-suited method for treating large field-cancerized skin areas.

In PDT a photosensitizing cream is applied on the skin and let to absorb. After absorption to the skin cells the photosensitizer changes into protoporphyrin IX (PpIX). PpIX reacts with visible light causing a phototoxic reaction which destroys cancer cells targetedly. After absorption the skin can be illuminated using a red lamp (conventional PDT) or natural daylight (NDL-PDT) as the absorption spectrum peaks of PpIX are within the visual spectrum of light.

In Finland the approved photosensitizers for PDT are methyl 5-aminolevulinate cream (MAL, Metvix®, Galderma) and aminolevulinic acid gel (BF-200 ALA, Ameluz®, Biofrontera AG). They both have been clinically studied and proved effective in conventional PDT but in NDL-PDT mainly MAL has been in focus of studies. To our knowledge there is only research report concerning the use of BF-200 ALA in NDL-PDT (Neittaanmaki-Perttu et al 2014) which is a study of our own research group. In this study BF-200 ALA appeared to be more effective than MAL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with widespread AK lesions symmetrically on face or scalp (at least 3 actinic keratoses symmetrically on face or scalp)
* AKs of grade I-II

Exclusion Criteria:

* Thick grade III AKs
* Previous treatment for actinic keratosis on the same skin area during preceding 6 months
* Porfyria or solar dermatitis
* Allergy for photosensitizers used in the study
* Pregnant or breastfeeding patients
* Impaired general condition (patient can't manage required 2 hours in sunlight outdoors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Clinical healing of actinic keratoses | 12 months
  Participant's AKs in the treatment areas are counted and categorized clinically in three grades I-III (Olsen et al. 1991) before the NDL-PDT treatment. The clinical healing of actinic keratoses will be assessed by a dermatologist 12 months after the treatment.

SECONDARY OUTCOMES:
Assessing pain experienced by participants: comparing the difference in symmetrical treatment areas of face or scalp | 1 day
  Participants will be asked to fill visual analogue scales (VAS) about pain experienced on both treatment sides of the face or scalp. Pain is assessed during the DL-PDT and after the treatment until the evening.

OTHER OUTCOMES:
Primary treatment reaction of skin | 1 week
  The participants will come to clinic 5-7 days after treatment and nurse will photograph both treatment sides. Primary treatment reaction of skin will be single-blindedly assessed from the photographs. A dermatologist will assess which side of the face or scalp presents a stronger reaction.
Dermatoecological analyses of the treatment costs | 12 months
  Researchers will analyze the cost-efficacy of the treatments using decision tree, sensitivity analysis, ICER and QALY-analyses to decide with treatment modality is more preferable. The differences in cost-efficacy will most likely depend on the light sensitizer costs and their efficacy on the treated lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Janne Rasanen, Lic. Med., Principal Investigator — Päijänne Tavastia Central Hospital; Mari Gronroos, D.Med.Sc., Study Director — Päijänne Tavastia Central Hospital; Noora Neittaanmaki-Perttu, D.Med.Sc., Study Chair — Helsinki University Central Hospital; Mari Salmivuori, Lic. Med., Study Chair — Päijänne Tavastia Central Hospital; Leea Ylitalo, D.Med.Sc., Study Chair — Tampere University Hospital; Johanna Hagman, D.Med.Sc., Study Chair — Vaasa Central Hospital, Vaasa, Finland; Ida Knutar, Lic. Med., Study Chair — Vaasa Central Hospital, Vaasa, Finland
Locations (3):
- Finland (3):
  - Päijät-Häme Central Hospital, Lahti
  - Tampere University Hospital, Tampere
  - Vaasa Central Hospital, Vaasa

REFERENCES:
- [Result] Rasanen JE, Neittaanmaki N, Ylitalo L, Hagman J, Rissanen P, Ylianttila L, Salmivuori M, Snellman E, Gronroos M. 5-aminolaevulinic acid nanoemulsion is more effective than methyl-5-aminolaevulinate in daylight photodynamic therapy for actinic keratosis: a nonsponsored randomized double-blind multicentre trial. Br J Dermatol. 2019 Aug;181(2):265-274. doi: 10.1111/bjd.17311. Epub 2019 Jan 2. PMID 30329163